CLINICAL TRIAL: NCT01717365
Title: SCOPE: A Psychometric Study
Brief Title: Psychometric / Validation Study
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Patricia Bowyer, Patricia Bowyer, EdD, , MS, OTR, FAOTA, Texas Woman's University
Other Study IDs: 15007
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: To Determine the Psychometric Properties of the Short Child Occupational Profile
Keywords: SCOPE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OTs: Occupational therapists

SUMMARY:
Data for the study will be collected from therapist across the world. The therapists will share data they have already compiled from their caseload. Data will be stripped of all personal identifiers and personal health information. The TWU SCOPE research team has no contact with clients whose assessment data is being shared for secondary analysis or clinical data repository. For educational and training purposes clients can be videotaped by the therapist who will obtain consent and/or assent from the client. Not every client will be videotaped. The subjects from the data shared by the therapists are from the ages of 0-21, both male and female, and of any ethnicity. The total amount of data collected from all participating therapists will be 500 pieces.

DETAILED DESCRIPTION:
Therapists will be recruited by a TWU SCOPE research team member via email. Therapists who wish to participate will send a data sharing letter to the PI of the study. Once the TWU SCOPE research team has received the data sharing letter, a clinical data packet will then be distributed to the therapist through the U.S. mail or an email will be sent containing a web address link to http://www.myweb.twu.edu/~ttioseco for access to the clinical data packet via the internet. Those therapists who collect ten pieces or more of de-identified data and send them to the TWU SCOPE research team will receive an incentive in the form of a gift card.

Flow Chart of Research Study Process Collaborators (share new de-identified data) → databank (new de-identified data input) → data analysis (analysis of new and old de-identified data) → publication/presentation

No risks are involved because data collected is without any personal identifiers.

ELIGIBILITY:
Inclusion Criteria:

Subjects receiving therapy from participating therapists.

Exclusion Criteria:

Age over 21.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The subjects from the data shared by the therapists are from the ages of 0-21, both male and female, and of any ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)

PRIMARY OUTCOMES:
To determine the psychometric properties of the Short Child Occupational Profile Validate SCOPE | 36 months
  To determine the psychometric properties of the Short Child Occupational Profile (SCOPE) and validate the SCOPE.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University, Houston, Texas, United States